CLINICAL TRIAL: NCT07027371
Title: Evaluation of Care Provided for Splenectomized Children and the Role of Patients' Education in Its Improvement
Brief Title: Post Splenectomy Care Assessment and the Role of Patient Education in Its Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Saad Nassim, Assistant Professor of Pediatrics, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MS-486-2021
Record Dates: First submitted 2025-06-04; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2021-04

CONDITIONS: Splenectomized Patients
Keywords: Overwhelming post splenectomy infections; splenectomy; chemoprophylaxis; vaccination; encapsulated organisms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional group (Experimental): Splenectomized patients above 15 years and caregivers of patients below 15 years received a questionnaire that included questions enquiring about age, gender, education level, disease type, duration of illness, age at splenectomy, duration since splenectomy, reception of preoperative vaccines, compliance to post splenectomy booster doses and penicillin prophylaxis, and the reasons for non-compliance if any, and their perception regarding red flags of Overwhelming Post Splenectomy Infection "OPSI". Based on the gaps of care identified in the essential questionnaire, educational material about perisplenectomy care was obtained. A knowledge test and a printed brochure were designed based on the knowledge script. Candidates who agreed to complete the study were asked to fill in individually the pre-education knowledge test. The brochures were then handed to each patient or caregiver. Participants were encouraged to read the brochure. Then they completed the post-education knowledge test
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Health education — Health education was given in the form of a printed colored brochure designed in easy-to-understand Arabic language. Participants were encouraged to read the brochure thoroughly and as many times as needed and to ask questions to the researchers if they had any.

SUMMARY:
The goal of this trial is to evaluate compliance to booster vaccines and chemoprophylaxis in children who underwent a splenectomy and to assess the knowledge regarding this aspect before and after giving education.

DETAILED DESCRIPTION:
The term "overwhelming post-splenectomy infection" (OPSI) refers to a rapid fatal syndrome occurring in individuals following removal of the spleen. OPSI can progress from a mild flu-like illness to fulminant sepsis in a short time period and has high mortality rate despite maximal treatment. The mainstays of infectious diseases prevention in asplenic subjects include: 1) patient and family education, 2) vaccinations, 3) prophylactic antimicrobial therapy in selected people, 4) early empirical antimicrobial therapy for febrile episodes, 5) early management of animal bites. Studies demonstrated that patients were neither compliant to postsplenectomy booster vaccines nor chemoprophylaxis with oral penicillin. Inadequate information and lack of sufficient education seem to be the major culprit behind this lack of awareness.

The study will be carried out at the Pediatric Hematology Clinic, Cairo University Children Hospital.

Candidates will be given questionnaires that will inquire about education level, disease type, age, duration of illness, age at splenectomy, duration of splenectomy , reception of preoperative vaccines (Pneumococcal, Hemophilus, Meningococcal vaccines) , compliance to postsplenectomy booster doses and penicillin prophylaxis , and if not what are the reasons for that.

Patients will also be given written information educating them about OPSI, its red flags and the importance of post splenectomy care. Interview questionnaire will be given to patients before and after education.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 15 years who had undergone splenectomy
* Caregivers of patients aged below 15 years who had undergone splenectomy

Exclusion Criteria:

* Illiterate candidates
* Candidates who refuse to take part in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Candidates' knowledge about the different aspects of post splenectomy hazards and methods of care | At baseline and immediately after intervention
  A questionnaire designed by the hematology team inquiring about different aspects of post splenectomy hazards and methods of care was handed to candidates. Each correct answer was given a score of 1. A score was summed up and a total score (as a percentage of correct answers) was given.

SECONDARY OUTCOMES:
To detect the rate of vaccination (defined as the percentage of people who have received vaccines) to pneumococcal, meningococcal and hemophilus influenza vaccine among the studied population (splenectomized patients). | At time of enrollment in the study
  This was achieved through a questionnaire inquiring about the reception of pneumococcal, meningococcal and hemophilus influenza vaccine among other data designed and given to candidates.
To detect the percentage of patients who received post splenectomy chemoprophylaxis among the studied population. | At time of enrollment in the study
  This was achieved through a questionnaire inquiring about the reception of chemoprophylaxis, handed to the candidates.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Faculty of Medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study are available from the investigator on reasonable request